CLINICAL TRIAL: NCT06450717
Title: Implementation of a Pilot Telerehabilitation Network in Pediatric Patients With Complex Neurodisabilities MedeaNeuroTelerehab-Net (MENTE.NET Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 850
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Neurological Diseases or Conditions
Keywords: Neurological condition; Telerehabilitation

STUDY DESIGN:
Intervention Model Description: The study is a two-year multicenter prospective clinical-experimental study. The project involves the initial small-scale application of a telerehabilitation study protocol to test whether the methodology is appropriate, establish its feasibility, and derive useful information for sample size calculation for subsequent randomized trials. For prospective data collection, patients will be consecutively enrolled at participating centers. At least 10 patients (age 4-18) per pole are expected to be enrolled in this pilot phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRRS group (Experimental): Participants will receive telerehabilitation treatment based delivered by Khymeia VRRS technology platform. The VRRS device, in the home version, is used in tele-rehabilitation mode. There are two modes of operation in tele-rehabilitation: on line mode: the therapist is able to take control of the system remotely and interact with the patient in real time through the integrated two-way video conferencing system with pan and zoom camera with which the VRRS is equipped; off-line mode: the therapist can prepare a list of exercises to be performed by the patient at home, assisted by the "smart virtual assistant" who guides the patient in the execution of the rehabilitation program. The home device automatically records all activities performed by the patient independently. The therapist can connect to the home device at any time to review the tests performed or modify the exercise list or make appropriate changes to the specific patient's rehabilitation program.
  Interventions: Device: Khymeia VRRS

INTERVENTIONS:
Device: Khymeia VRRS — VRRS is an electronic device for remote rehabilitation of cognitive (e.g., memory, attention, spatial perception, logical-mathematical skills, language, executive functions...) and motor (gross and fine motor skills) functions. It can be used in on-line and off-line mode at home, and the exercises are chosen by the therapist according to the patient's specific difficulties and needs from a cognitive and motor library.
  Other Names: VRRS

SUMMARY:
This pilot study aims at networking the experience gained in neurorehabilitation of developmental neurodisabilities from the 3 poles of IRCCS Medea (Brindisi, Bosisio Parini, and Conegliano) to assess the feasibility of performing home-based telerehabilitation on cognitive and motor aspects through the Khymeia Virtual Reality Rehabilitation System (VRRS) platform.

DETAILED DESCRIPTION:
Few studies report the efficacy of telerehabilitation treatments in developmental age. The results suggest that it could be a promising tool for neurorehabilitation.The present pilot study aims at networking the experience gained in neurorehabilitation of developmental neurodisabilities from the 3 poles of IRCCS Medea (Brindisi, Bosisio Parini, and Conegliano) to evaluate the feasibility of performing home-based TR on cognitive and motor aspects through the Khymeia VRRS platform. VRRS represents an innovative system for immersive and non-immersive virtual reality rehabilitation and telerehabilitation.

In view of recent developments in Information and Communication Technologies (ICT) and their applicability to the neurological evaluation and rehabilitation context, VRRS instrumentation may represent a suitable methodology to assess the feasibility of a rehabilitation and telerehabilitation protocol for patients with complex neurodisabilities in pediatric age.

The present pilot project involves the use of the VRRS technology platform and the use of exercises performed in a 3D virtual and non-3D virtual environment. Implementation in the virtual environment of the exercises allows the therapist to set up, graduate, and modulate the selected exercises in the platform. The playful aspects and continuous performance monitoring and evaluation are then a key aspect in the rehabilitation process, as they keep the patient's motivation high. Through Home Tablets delivered to the patient, the platform makes possible home telerehabilitation through the proposal of cognitive and motor activities in 2 modes, Online (in the presence of the therapist) and Offline.

In order to test the feasibility of cognitive-motor rehabilitation intervention protocols carried out through VRRS, 30 patients (10 per research center) will be recruited and treated by using the VRRS library exercises. The VRRS exercises will be chosen according to the specific rehabilitation needs of each participant.

The study is designed as a two-year multicenter prospective clinical-experimental pilot study. The project involves the initial small-scale application of a telerehabilitation study protocol to test whether the methodology is appropriate, establish its feasibility, and derive useful information for sample size calculation for subsequent randomized trials. For prospective data collection, patients will be consecutively enrolled at participating centers.

If the VRRS is confirmed to be a suitable tool for conducting cognitive and motor TR in this clinical population as well, the present study may set the stage for future efficacy studies.

Other objectives of the study are:

* to identify within the network telerehabilitation programs aimed at improving cognitive and motor functions in developmental-age individuals with neurodisabilities, identifying common modes of intervention;
* to collect a longitudinal data set through the use of specific assessment batteries on motor, cognitive and functional adaptation functions, including from the perspective of ICF, secondary complications, autonomy, participation and quality of life. As a pilot study, conduct initial analyses of the effectiveness of interventions in order to create useful data for sample size calculation for subsequent randomized trials;
* to provide health policy makers with better scientific evidence on telerehabilitation in order to plan interventions aimed at better utilization and enhancement of these methods;
* to highlight good practices related to telerehabilitation by proposing a series of evaluations and recommendations aimed at fostering further improvement in the quality of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* congenital or acquired, cognitive or motor neurodisability;
* cooperation and abiity to understand the offered activities;
* where necessary, parents or legal guardians able to commit to and cooperate in a home-based telerehabilitation program.

Exclusion Criteria:

* Developmental disorders;
* Psychiatric disorders.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-06-09 (Actual); Study Completion 2024-06-09 (Actual)

PRIMARY OUTCOMES:
True or False? (VRRS Task - executive functioning) | baseline (immediately pre-training)
  The task requires the participant to answer true or false to statements that describe the mug design on the screen. As you advance in level, the features to be considered increase (e.g., color, number of objects, presence or absence of certain objects, etc.). The test aims to assess observation skills, comprehension and working memory. The test lasts 5 minutes and you will pass the level after 4 consecutive correct answers. The correctness of the answers and the number of total repetitions made are evaluated. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in individual performance pre- and post-intervention.
True or False? (VRRS Task - executive functioning) | post-training (approximatively at week 4)
  The task requires the participant to answer true or false to statements that describe the mug design on the screen. As you advance in level, the features to be considered increase (e.g., color, number of objects, presence or absence of certain objects, etc.). The test aims to assess observation skills, comprehension and working memory. The test lasts 5 minutes and you will pass the level after 4 consecutive correct answers. The correctness of the answers and the number of total repetitions made are evaluated. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in individual performance pre- and post-intervention.
Bells Test | baseline (immediately pre-training)
  This is a cancellation task and it gives a measure of visual selective attention. It requires participants to mark all the bells in 4 consecutives sheets. It gives both a measure of rapidity and accuracy. The task consists of 4 parts (4 visual research sheets presented in succession). For each of them there is a maximum time of 120 seconds. The accuracy score corresponds to the total number of bells found in the 120 seconds for each sheet. The quickness score corresponds to the total number of bells found in the first 30 seconds for each sheet. For both accuracy and rapidity scores, the z score ((score-average)/standard deviation) is calculated. A score below z= -2 indicates a poor performance.
Bells Test | post-training (approximatively at week 4)
  This is a cancellation task and it gives a measure of visual selective attention. It requires participants to mark all the bells in 4 consecutives sheets. It gives both a measure of rapidity and accuracy. The task consists of 4 parts (4 visual research sheets presented in succession). For each of them there is a maximum time of 120 seconds. The accuracy score corresponds to the total number of bells found in the 120 seconds for each sheet. The quickness score corresponds to the total number of bells found in the first 30 seconds for each sheet. For both accuracy and rapidity scores, the z score ((score-average)/standard deviation) is calculated. A score below z= -2 indicates a poor performance.
Visual attention (NEPSY II task) | baseline (immediately pre-training)
  This is a cancellation task and it gives a measure of visual selective attention. It requires participants to mark all faces corresponding to the target faces printed on two sheets among similar faces (distractors). The allotted time is 180 seconds. The raw score is converted to a standard score. Standard scores between 8 and 12 are within the normal range. They turn out to be lower than expected when less than 8.
Visual attention (NEPSY II task) | post-training (approximatively at week 4)
  This is a cancellation task and it gives a measure of visual selective attention. It requires participants to mark all faces corresponding to the target faces printed on two sheets among similar faces (distractors). The allotted time is 180 seconds. The raw score is converted to a standard score. Standard scores between 8 and 12 are within the normal range. They turn out to be lower than expected when less than 8.
Attention and concentration software (exercise 3) | baseline (immediately pre-training)
  The test requires a computer and includes three different exercises that measure auditory, visual and spatial attention, respectively. It gives a measure of rapidity and accuracy for each type of exercise. There is no advancement level, it is administered at level 1 only. Tables are available for all the tests in this CD that allow you to see the reference percentile (for errors) and to calculate the z-point (for the velocity dimension). Each table shows the number of errors that corresponds to the lowest quartile (25%). A number of errors exceeding this score is considered an indication of poor performance. Regarding speed, the tables report averages and standard deviations and allow calculation of the z-point. As above scores below z -2 indicate poor performance.
Attention and concentration software (exercise 3) | post-training (approximatively at week 4)
  The test requires a computer and includes three different exercises that measure auditory, visual and spatial attention, respectively. It gives a measure of rapidity and accuracy for each type of exercise. There is no advancement level, it is administered at level 1 only. Tables are available for all the tests in this CD that allow you to see the reference percentile (for errors) and to calculate the z-point (for the velocity dimension). Each table shows the number of errors that corresponds to the lowest quartile (25%). A number of errors exceeding this score is considered an indication of poor performance. Regarding speed, the tables report averages and standard deviations and allow calculation of the z-point. As above scores below z -2 indicate poor performance.
Melbourne Assessment of Unilateral Upper Limb Function | baseline (immediately pre-training)
  MA2 evaluates 4 elements (Range of movement, Accuracy of reach and placement, Dexterity of grasp, release and manipulation, and Fluency of movement) of upper limb movement quality in children (2.5-15 y.o.) with a neurological impairment. The full test requires the child to reach to, grasp, release and manipulate simple objects, and each performance is video recorded. Scoring is completed across the 30 score items using a 3, 4 or 5-point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale. A final score is reported as 4 separate scores (one for each element measured). A raw score for each sub-scale is converted to a percentage of the maximum possible score for that sub-scale. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.
Melbourne Assessment of Unilateral Upper Limb Function | post-training (approximatively at week 3)
  MA2 evaluates 4 elements (Range of movement, Accuracy of reach and placement, Dexterity of grasp, release and manipulation, and Fluency of movement) of upper limb movement quality in children (2.5-15 y.o.) with a neurological impairment. The full test requires the child to reach to, grasp, release and manipulate simple objects, and each performance is video recorded. Scoring is completed across the 30 score items using a 3, 4 or 5-point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale. A final score is reported as 4 separate scores (one for each element measured). A raw score for each sub-scale is converted to a percentage of the maximum possible score for that sub-scale. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.
Melbourne Assessment of Unilateral Upper Limb Function | follow up (approximatively 1 month post-training)
  MA2 evaluates 4 elements (Range of movement, Accuracy of reach and placement, Dexterity of grasp, release and manipulation, and Fluency of movement) of upper limb movement quality in children (2.5-15 y.o.) with a neurological impairment. The full test requires the child to reach to, grasp, release and manipulate simple objects, and each performance is video recorded. Scoring is completed across the 30 score items using a 3, 4 or 5-point scale and individually defined scoring criteria. Item scores relating to each element of movement measured are summed within the corresponding sub-scale. A final score is reported as 4 separate scores (one for each element measured). A raw score for each sub-scale is converted to a percentage of the maximum possible score for that sub-scale. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.
Scala Besta | baseline (immediately pre-training)
  The Besta scale evaluates hand grip on request with standard material (1.5-3.5 cm dice), spontaneous use with game material that implies bimanuality and spontaneous use of the hand in praxis activities (with proposals for independent activities such as feeding, cleaning, clothing). The assessment is intended for use with children aged 6 to 12 years. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in individual's performance pre- and post-intervention.
Scala Besta | post-training (approximatively at week 3)
  The Besta scale evaluates hand grip on request with standard material (1.5-3.5 cm dice), spontaneous use with game material that implies bimanuality and spontaneous use of the hand in praxis activities (with proposals for independent activities such as feeding, cleaning, clothing). The assessment is intended for use with children aged 6 to 12 years. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in individual's performance pre- and post-intervention.
Scala Besta | follow up (approximatively 1 month post-training)
  The Besta scale evaluates hand grip on request with standard material (1.5-3.5 cm dice), spontaneous use with game material that implies bimanuality and spontaneous use of the hand in praxis activities (with proposals for independent activities such as feeding, cleaning, clothing). The assessment is intended for use with children aged 6 to 12 years. There are no cutoff points. However, raw scores can be statistically analyzed for evaluation changes in individual's performance pre- and post-intervention.
Movement Assessment Battery for Children (M-ABC)-II | baseline (immediately pre-training)
  The M-ABC was specifically developed for identifying and evaluating children with mild to moderate motor impairment. The test is divided into three age groups (3-6; 7-10; 11-16). For each age group, eight tasks are provided, grouped into three sections: manual dexterity, aiming and catching, and balance. Raw scores for each of the tasks and for each age group can be converted into standard scores (with a mean of 10 and a standard deviation of 3) and percentiles. A standard score equivalent to the 5th percentile is considered pathological. In our study, we will administer the same test evaluating manual dexterity to all subjects (regardless of age) and analyze the changes in raw scores between pre- and post-intervention.
Movement Assessment Battery for Children (M-ABC)-II | post-training (approximatively at week 3)
  The M-ABC was specifically developed for identifying and evaluating children with mild to moderate motor impairment. The test is divided into three age groups (3-6; 7-10; 11-16). For each age group, eight tasks are provided, grouped into three sections: manual dexterity, aiming and catching, and balance. Raw scores for each of the tasks and for each age group can be converted into standard scores (with a mean of 10 and a standard deviation of 3) and percentiles. A standard score equivalent to the 5th percentile is considered pathological. In our study, we will administer the same test evaluating manual dexterity to all subjects (regardless of age) and analyze the changes in raw scores between pre- and post-intervention.
Movement Assessment Battery for Children (M-ABC)-II | follow up (approximatively 1 month post-training)
  The M-ABC was specifically developed for identifying and evaluating children with mild to moderate motor impairment. The test is divided into three age groups (3-6; 7-10; 11-16). For each age group, eight tasks are provided, grouped into three sections: manual dexterity, aiming and catching, and balance. Raw scores for each of the tasks and for each age group can be converted into standard scores (with a mean of 10 and a standard deviation of 3) and percentiles. A standard score equivalent to the 5th percentile is considered pathological. In our study, we will administer the same test evaluating manual dexterity to all subjects (regardless of age) and analyze the changes in raw scores between pre- and post-intervention.
System Usability Scale (SUS) for PCI | baseline (immediately pre-training)
  SUS is a quick and dirty survey scale that assess the usability of a give product or service. It is composed of 10 statements that are scored on a 5-point scale of strength of agreement. Final score for the SUS can range from 0 to 100, where higher scores indicate better usability. A product with a score greater than 70 indicates a product with good usability.
System Usability Scale (SUS) for SMA | post-training (approximatively at week 3)
  SUS is a quick and dirty survey scale that assess the usability of a give product or service. It is composed of 10 statements that are scored on a 5-point scale of strength of agreement. Final score for the SUS can range from 0 to 100, where higher scores indicate better usability. A product with a score greater than 70 indicates a product with good usability.
Revised Hammersmith Scale (RHS) | baseline (immediately pre-training)
  The RHS is a clinician rated SMA specific outcome measure containing 36 items which assess physical motor performance. The scale assesses motor functional activities related to sitting, supine, rolling, prone, ability to move and get up from the floor, balance, standing, run/ walk, stairs, ascending and descending a step and the ability to jump. Thirty-three items are graded according to an ordinal 0, 1, 2 scale where 0 represents the least physical ability or function achieved, and 2 the highest. Three items are graded 0 and 1 where 0 represents an inability to complete the item, and 1 represents achieving the item. There are no cutoff points. However, scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.
Revised Hammersmith Scale (RHS) | post-training (approximatively at week 3)
  The RHS is a clinician rated SMA specific outcome measure containing 36 items which assess physical motor performance. The scale assesses motor functional activities related to sitting, supine, rolling, prone, ability to move and get up from the floor, balance, standing, run/ walk, stairs, ascending and descending a step and the ability to jump. Thirty-three items are graded according to an ordinal 0, 1, 2 scale where 0 represents the least physical ability or function achieved, and 2 the highest. Three items are graded 0 and 1 where 0 represents an inability to complete the item, and 1 represents achieving the item. There are no cutoff points. However, scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.
Revised Upper Limb Module (RULM) Scale | baseline (immediately pre-training)
  The scale consists of an entry item to establish functional levels and 19 items covering distal to proximal movements. The entry item is a modified version of the Brooke scale, including activities ranging from no functional use of hands (score 0) to full bilateral shoulder abduction (score 6). The entry item does not contribute to the total score but serves as a functional classification of overall upper limb functional ability. Of the remaining 19 items, 18 are scoredon a 3 point scoring system and 1 item is scored on a 2 point scoring system. The total score ranges from 0, if all the items cannot be performed, to 37, if all the activities are achieved fullywithout any compensation. There are no cutoff points. However, scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.
Revised Upper Limb Module (RULM) Scale | post-training (approximatively at week 3)
  The scale consists of an entry item to establish functional levels and 19 items covering distal to proximal movements. The entry item is a modified version of the Brooke scale, including activities ranging from no functional use of hands (score 0) to full bilateral shoulder abduction (score 6). The entry item does not contribute to the total score but serves as a functional classification of overall upper limb functional ability. Of the remaining 19 items, 18 are scoredon a 3 point scoring system and 1 item is scored on a 2 point scoring system. The total score ranges from 0, if all the items cannot be performed, to 37, if all the activities are achieved fullywithout any compensation. There are no cutoff points. However, scores can be statistically analyzed for evaluation changes in an individual's performance pre- and post-intervention.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventor (PedsQLTM) for PCI | baseline (immediately pre-training)
  PedsQLTM is the standard generic core scale of quality of life (QoL) to measure the physical and psychosocial health of either healthy or ill children. The PedsQL includes 23 questions with a five-point rating scale (range of 0 to 4 points based on the agreement in each statement). Questions cover the following areas: physical health and psychosocial health, including emotional, social, and cognitive/school functioning. The scores were transformed into full scores of a maximum of 100 points in each area: 100 points meant good QoL, while 0 points meant QoL with very frequent problems. The reliability and validity of PedsQL generic core scales have been well established in healthy and sick populations. There are no cutoff points to distinguish high QoL from low QoL. However, the scores can be statistically analyzed longitudinally to evaluate a change in quality of life following an intervention.
Pediatric Quality of Life Inventor (PedsQLTM) for PCI | post-training (approximatively at week 3)
  PedsQLTM is a standard generic core scale of quality of life (QoL) to measure the physical and psychosocial health of either healthy or ill children. The PedsQL includes 23 questions with a five-point rating scale (range of 0 to 4 points based on the agreement in each statement). Questions cover the following areas: physical health and psychosocial health, including emotional, social, and cognitive/school functioning. The scores were transformed into full scores of a maximum of 100 points in each area: 100 points meant good QoL, while 0 points meant QoL with very frequent problems. The reliability and validity of PedsQL generic core scales have been well established in healthy and sick populations. There are no cutoff points to distinguish high QoL from low QoL. However, the scores can be statistically analyzed longitudinally to evaluate a change in quality of life following an intervention.
Pediatric Quality of Life Inventor (PedsQLTM) for PCI | follow up (approximatively 1 month post-training)
  PedsQLTM is a standard generic core scale of quality of life (QoL) to measure the physical and psychosocial health of either healthy or ill children. The PedsQL includes 23 questions with a five-point rating scale (range of 0 to 4 points based on the agreement in each statement). Questions cover the following areas: physical health and psychosocial health, including emotional, social, and cognitive/school functioning. The scores were transformed into full scores of a maximum of 100 points in each area: 100 points meant good QoL, while 0 points meant QoL with very frequent problems. The reliability and validity of PedsQL generic core scales have been well established in healthy and sick populations. There are no cutoff points to distinguish high QoL from low QoL. However, the scores can be statistically analyzed longitudinally to evaluate a change in quality of life following an intervention.
Pediatric Quality of Life Inventor (PedsQLTM) for SMA | baseline (immediately pre-training)
  PedsQLTM is a standard generic core scale of quality of life (QoL) to measure the physical and psychosocial health of either healthy or ill children. The PedsQL includes 23 questions with a five-point rating scale (range of 0 to 4 points based on the agreement in each statement). Questions cover the following areas: physical health and psychosocial health, including emotional, social, and cognitive/school functioning. The scores were transformed into full scores of a maximum of 100 points in each area: 100 points meant good QoL, while 0 points meant QoL with very frequent problems. The reliability and validity of PedsQL generic core scales have been well established in healthy and sick populations. There are no cutoff points to distinguish high QoL from low QoL. However, the scores can be statistically analyzed longitudinally to evaluate a change in quality of life following an intervention.
Pediatric Quality of Life Inventor (PedsQLTM) for SMA | post-training (approximatively at week 3)
  PedsQLTM is a standard generic core scale of quality of life (QoL) to measure the physical and psychosocial health of either healthy or ill children. The PedsQL includes 23 questions with a five-point rating scale (range of 0 to 4 points based on the agreement in each statement). Questions cover the following areas: physical health and psychosocial health, including emotional, social, and cognitive/school functioning. The scores were transformed into full scores of a maximum of 100 points in each area: 100 points meant good QoL, while 0 points meant QoL with very frequent problems. The reliability and validity of PedsQL generic core scales have been well established in healthy and sick populations. There are no cutoff points to distinguish high QoL from low QoL. However, the scores can be statistically analyzed longitudinally to evaluate a change in quality of life following an intervention.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Alessandra Bardoni, Bosisio Parini, Lecco
  - Andrea Martinuzzi, Conegliano, Treviso
  - Antonio Trabacca, Brindisi